CLINICAL TRIAL: NCT00003929
Title: Combined Modality Therapy of AIDS-Related and Immunocompetent Primary CNS Lymphoma (PCL) Using Filgrastim (G-CSF)
Brief Title: Chemotherapy, Filgrastim, and Radiation Therapy in Treating Patients With Primary Central Nervous System Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU3496; P30CA043703 (NIH); CWRU-3496 (Other: Case Comprehensive Cancer Center); CWRU-AMC-2A-93; NCI-G99-1533
Record Dates: First submitted 1999-11-01; First posted 2004-07-26 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma
Keywords: primary central nervous system lymphoma; AIDS-related primary CNS lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Filgrastim; Lomustine; Procarbazine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — Filgrastim (G-CSF) is administered subcutaneously daily on days 12-21 and days 33-42, until absolute neutrophil counts recover. Patients with a complete response after 6 weeks receive one additional course of chemotherapy prior to radiotherapy.
Drug: lomustine — Oral lomustine on day 1. Patients with a complete response after 6 weeks receive one additional course of chemotherapy prior to radiotherapy.
Drug: procarbazine hydrochloride — Oral procarbazine on days 1-10 and days 22-31. Patients with a complete response after 6 weeks receive one additional course of chemotherapy prior to radiotherapy.
Radiation: radiation therapy — Whole brain radiotherapy is administered daily for 28 days beginning 1-3 weeks following chemotherapy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy with radiation therapy may kill more cancer cells. Colony-stimulating factors such as filgrastim allow doctors to give higher doses of chemotherapy drugs to kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of lomustine, procarbazine, filgrastim, and radiation therapy in treating patients who have primary central nervous system lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine response rate, response duration, and survival of patients with AIDS-related or immunocompetent primary central nervous system lymphoma after treatment with oral lomustine and procarbazine, filgrastim (G-CSF), and radiotherapy. II. Determine toxicity of this combined modality in these patients. III. Determine quality of life of these patients.

OUTLINE: Patients are stratified by CD4 count (50/mm3 and under vs greater than 50/mm3). Patients receive oral lomustine on day 1 and oral procarbazine on days 1-10 and days 22-31. Filgrastim (G-CSF) is administered subcutaneously daily on days 12-21 and days 33-42, until absolute neutrophil counts recover. Patients with a complete response after 6 weeks receive one additional course of chemotherapy prior to radiotherapy. Patients with a partial response, stable disease, or disease progression after 6 weeks proceed to radiotherapy without receiving a second course of chemotherapy. Whole brain radiotherapy is administered daily for 28 days beginning 1-3 weeks following chemotherapy. Quality of life is assessed prior to therapy, at 3 and 6 weeks, and then every 2 months following radiotherapy. Patients are followed every 2 months until death.

PROJECTED ACCRUAL: Approximately 16 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven AIDS-related non-Hodgkin's lymphoma of the CNS or non AIDS-related,non-Hodgkin's lymphoma of CNS also eligible, if not eligible for higher priority clinical trial

PATIENT CHARACTERISTICS: Age: 0-120 Performance status: ECOG 0-2 Life expectancy: At least 6 weeks Hematopoietic: WBC at least 1500/ mm3 Platelets at least 50,000/mm3 Hepatic: Serum bilirubin no greater than 3.0 mg/dL Renal: Serum creatinine no greater than 3.0 mg/dL Cardiovascular: Pulmonary: Other: Active infection(s) allowed if drug receiving treatment No Zidovudine during combined modality chemotherapy and radition Negative CSF cytology

PRIOR CONCURRENT THERAPY: Biologic therapy: Chemotherapy: No prior chemotherapy Endocrine therapy: Steroids may be used concurrently. Doses should be as low as possible. Increases in steroids above study's upper limit will result in patient going off study. Radiotherapy: No prior radiotherapy Surgery: Prior surgical debulking allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-06; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness of lomustine, procarbazine, filgrastim, and radiation therapy in treating patients who have primary central nervous system lymphoma. | Patients with a CR after 6 weeks receive one additional course of chemotherapy prior to radiotherapy. Patients with a PR, stable disease, or disease progression after 6 weeks proceed to radiotherapy without receiving a second course of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States